CLINICAL TRIAL: NCT00720356
Title: A Phase II Study of Bevacizumab and Erlotinib After Radiation Therapy and Temozolomide in Patients With Newly Diagnosed Glioblastoma Without MGMT Promoter Methylation
Brief Title: Bevacizumab and Erlotinib After Radiation Therapy and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma Multiforme or Gliosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Jeffrey Raizer, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 07C3; NU 07C3 (Other: Northwestern University); BTTC08-01 (Other: U.T. M.D. Anderson Cancer Center); STU00002792 (Other: Northwestern University IRB)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): erlotinib and bevacizumab
  Interventions: Drug: bevacizumab; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: bevacizumab — 10mg/kg administered intravenously every 2 weeks
  Other Names: Avastin
Drug: erlotinib hydrochloride — 150 mg/daily orally
  Other Names: erlotinib; CP-358, 774; Tarceva

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving bevacizumab together with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with erlotinib works after radiation therapy and temozolomide in treating patients with newly diagnosed glioblastoma multiforme or gliosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall survival of patients with newly diagnosed glioblastoma multiforme (GBM) with unmethylated MGMT promoter treated with bevacizumab and erlotinib hydrochloride after radiotherapy and temozolomide.

Secondary

* To determine the 12- and 24-month progression-free survival (PFS) of patients with newly diagnosed GBM with unmethylated MGMT promoter treated with this regimen.
* To assess radiographic response rates.
* To perform correlative tissue assays.
* To collect safety data on the combination of bevacizumab and erlotinib hydrochloride in patients with newly diagnosed GBM with unmethylated MGMT promoter treated with bevacizumab and erlotinib hydrochloride after radiotherapy and temozolomide.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy (either intensity-modulated radiation therapy or 3-D conformal radiotherapy) once daily 5 days a week and receive oral temozolomide concurrently with radiotherapy once daily for 6 weeks (as planned). Patients whose tumor has a methylated MGMT promoter are removed from study.

Approximately 4 weeks after completion of radiotherapy and temozolomide, patients receive bevacizumab IV over 30-90 minutes on days 1 and 15 and oral erlotinib hydrochloride once daily on days 1-28. Treatment with bevacizumab and erlotinib hydrochloride repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at approximately 30 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed glioblastoma multiforme (GBM) or gliosarcoma
* Undergoing or plan to undergo treatment with radiotherapy and concurrent temozolomide for 6 weeks
* Unmethylated MGMT promoter status must be determined before completing radiotherapy

  * Tumor must be MGMT negative to receive bevacizumab and erlotinib hydrochloride
* Patients who are post biopsy or tumor resection allowed provided a post-operative MRI is done no more than 96 hours after surgery (in order for an accurate assessment to be done post radiotherapy):

  * Evaluable or measurable disease after resection of recurrent tumor is not mandated for eligibility
* Patients who started radiotherapy and temozolomide prior to study entry are eligible as long as the gene methylation status is determined before starting bevacizumab and erlotinib hydrochloride

  * Radiotherapy plans need to be verified to confirm the treatment plan meets the study requirement based on the PI assessment
  * No progressive disease based on MRI or CT scan per the investigators assessment

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy > 12 weeks
* WBC > 3,000/μL
* ANC > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 10 g/dL
* SGOT/SGPT < 3 times upper limit of normal (ULN)
* Bilirubin < 3 times ULN
* Creatinine < 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No significant medical illness that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to tolerate this therapy, or any disease that will obscure toxicity or dangerously alter drug metabolism
* No proteinuria at screening, as demonstrated by either of the following:

  * Urine protein:creatinine (UPC) ratio < 1.0
  * Urine dipstick for proteinuria < 2+ OR ≤ 1g protein by 24-hour urine collection
* No inadequately controlled hypertension (defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 100 mm Hg) on antihypertensive medications
* No history of hypertensive crisis or hypertensive encephalopathy
* No New York Heart Association class II-IV congestive heart failure
* No history of myocardial infarction or unstable angina within 6 months prior to study enrollment
* No history of stroke or transient ischemic attack within 6 months of study enrollment
* No symptomatic peripheral vascular disease
* No significant vascular disease (i.e., aortic aneurysm or aortic dissection)
* No evidence of bleeding diathesis or coagulopathy
* No significant traumatic injury within 28 days prior to study enrollment
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* No serious, nonhealing wound, ulcer, or bone fracture
* No known HIV positivity

  * HIV testing is not required for study participation
* No history of any other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years

PRIOR CONCURRENT THERAPY:

* No chemotherapy is allowed prior to starting radiotherapy and temozolomide, including polifeprosan 20 with carmustine implant (Gliadel wafers)
* No major surgical procedure or open biopsy within 28 days prior to study enrollment or the anticipation of need for major surgical procedure during the course of the study
* No core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* Concurrent nonenzyme-inducing anticonvulsants allowed

  * More than 2 weeks (before starting erlotinib hydrochloride and bevacizumab) since prior and no concurrent enzyme-inducing anticonvulsant
* No other concurrent experimental agents
* Not concurrently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-07-07 (Actual); Primary Completion 2014-06-24 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Raizer, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Northwestern University, Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Neuro-Oncology Associates at Baylor University Medical Center, Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - The Methodist Hospital Neurological Institute, Houston, Texas
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was ready for accrual March 12, 2009 with an accrual goal of up to 50 patients. The first patient was enrolled on July 7 2009. Accrual was suspended on July 29 2010 and reopened on March 30, 2011. The study was closed permanently on November 03, 2011 with an accrual of 48 patients treated on study after screening 115 patients.
Pre-assignment Details: Registration is a two step process. ICF signed, tissue sent off and MGMT promoter methylation status determined eligibility. Patients with unmethylated MGMT promoters will be complete the second registration step and be treated on study. Patients with methylated MGMT promoters will not be treated on study.
Groups:
- Erlotinib and Bevacizumab Combination Treatment: Erlotinib and bevacizumab
  Bevacizumab: 10mg/kg administered intravenously every 2 weeks
  Erlotinib hydrochloride: 150 mg/daily orally
Period: Registration to Study
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Started | 115
Completed Registration Step 1 | 115
Completed Registration Step 2 | 48
Completed | 48
Not Completed | 67
Not completed — Determined to have methylated MGMT | 67
Period: Reached 1st Response/2 Cycles
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Started | 48
Completed | 46
Not Completed | 2
Not completed — Progressive Disease | 1
Not completed — Withdrawal by Subject | 1
Period: Went on to be Treated Cycle 3
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Started | 46
Completed | 44
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Period: Follow up Until Death
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Started | 48 (All patients that are treated on study go into the follow up period)
Completed | 43
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Alive at last data collection | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 109
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 115
Methylated/unmethylated MGMT promoter [Count of Participants; unit: Participants] — After registration step 1 was completed, patients tissue was sent out for methylation MGMT determination. Only patients with unmethylated MGMT promoters were eligible for the study and completed registration step 2.
  Participants
    Methylated MGMT promoter | 67
    Unmethylated MGMT promoter | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) will be measured from the start of treatment until death from any cause. At data cut off patients remaining alive will be censored at the last known date of contact.
Time Frame: From start of treatment, during treatment and every 3 months following the end of treatment until death. Median follow up at time of OS data was 33 months.
Population: 2 patients were not evaluable - 1 patient withdrew consent and 1 patient completed less than 1 cycle of treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
Months | 13.2 [10.8 to 19.6]

2. Secondary Outcome: Progression-free Survival at 12 Months
Description: Progression free survival (PFS) will be assessed by CT or MRI scan using McDonald criteria. Progressive disease (PD) is defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). Stable or increased dose of steroids. PFS will be measured from the start of treatment until first documentation of PD or death.
Time Frame: At 12 months from start of treatment
Population: Two patients were determined not to be evaluable (one patient withdrew consent from the study and one patient completed one cycle)
Measure: Number; unit: percentage of patients
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
percentage of patients | 32

3. Secondary Outcome: Response Rate (RR)
Description: Response Rate (RR) will be defined as the best response seen during treatment measured by CT/MRI scan every 8 weeks during treatment using McDonald Criteria.
  CR=Complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients off steroids.
  PR=Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions. Stable/decreased dose of steroids.
  Stable/No Response=Does not qualify for CR, PR, or progression. The designation of Stable/No Response requires a minimum of 8 weeks duration. Stable/decreased dose of steroids.
  Progressive disease = 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease), worsening of evaluable disease, new lesions/site, failure to return for evaluation due to death or deteriorating condition.
Time Frame: From the start of treatment, every 2 cycles (1 cycle = 28 days) during treatment until progressive disease
Population: Two patients were determined not to be evaluable (one patient withdrew consent from the study and one patient complete one cycle of treatment only)
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
Participants
  Complete Response | 4
  Partial Response | 12
  Stable/no response | 28
  Progressive Disease | 0
  No Evaluable Disease (NED) | 2

4. Secondary Outcome: Safety of the Combination of Erlotinib and Bevacizumab in This Patient Population
Description: Toxicity data for combination treatment of erlotinib and bevacizumab will be collected on day 1 of every cycle (1 cycle = 28 days) during treatment according to the National Cancer Institute's Common Toxicity Criteria for adverse events version 3.0 (CTCAE v3.0). In general adverse events (AEs) will be graded according to the following:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: From the start of treatment, at the beginning of every cycle (1 cycle = 28 days) during treatment until 30 days after completion of treatment for up to 49 cycles.
Population: All patients that received at least one dose of study drug were evaluable for toxicity. Data for grade 3 and 4 toxicities during treatment were collected.
Measure: Number; unit: patients
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 48
patients
  Hyberbilirubinemia | 1
  Cerebrovascular ischemia | 1
  Dehydration | 1
  Dermatology/Skin | 1
  Hypertension | 3
  Fatigue | 3
  Leukocytes | 1
  Lymphopenia | 12
  Heartburn | 1
  Pain (not otherwise specified) | 1
  Pain abdomen | 1
  Pain head/headache | 1
  Bowel perforation | 1
  Hypophosphatemia | 1
  Rash/desqyamation | 5
  Rash/acneform | 2
  Syncope | 1
  Thrombosis/embolism | 2
  Wound complication | 1

5. Secondary Outcome: Progression Free Survival at 18 Months
Description: as for outcome 2
Time Frame: At 18 months from start of treatment
Population: Most patients had progressed before the 18 month time point. Data was not collected for PFS at 18 months.
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Changes in Tumor Blood Flow Based on MR Perfusion
Description: Data from consenting patients will be used to assess of changes in tumor blood flow based on MR perfusion using MRI scans. Two scans will be completed prior to treatment on study; the first after surgery buta before radiation, the second within 14 days before starting combination treatment or erlotinib and bevacizumab. Then scans will be completed every 2 cycles during treatment, where one cycle equals 28 days.
Time Frame: Prior to study treatment (after surgery, but before radiation), just before study treatment (within 14 days prior to first treatment) and then every 2 cycles during study treatment, where 1 cycle equals 28 days for a maximum of 49 cycles.
Population: This was an optional portion of the study that patients could participate in. Data was not collected or analyzed for this outcome measure.
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Gene Methylation Studies (Optional)
Description: Tissue and plasma collected from consenting patients in the study will be used to correlate tumor tissue with imaging and outcomes. Tissue will be collected before treatment on study begins and plasma will be collected the first day of treatment (before treatment) and every odd cycle after that, whilst on study treatment. Tissue and plasma analysis will be correlated with patients imaging results and response to to treatment
Time Frame: At baseline and then plasma only will be collected every odd cycle (1 cycle = 28 days) during treatment for a maximum of 49 cycles.
Population: This was an optional portion of the study for consenting patients. No data was collected and analyzed for this outcome measure.
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 0

8. Post Hoc Outcome: Progression Free Survival at 6 Months
Description: as for outcome 2
Time Frame: At 6 months from start of treatment
Population: Two patients were not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
percentage of patients | 66.3

9. Post Hoc Outcome: Overall Survival at 12 Months
Description: Overall Survival (OS) is measured from start of treatment until death from any cause.
Time Frame: At 12 months from start of treatment
Population: Two patients were not evaluable
Measure: Number; unit: percentage of patients
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
percentage of patients | 54.5

10. Post Hoc Outcome: Overall Survival at 24 Months
Description: Overall Survival (OS) will be measured from start of treatment until death of any cause
Time Frame: At 24 months from first treatment
Population: Two patients were not evaluable
Measure: Number; unit: percentage of patients
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
percentage of patients | 32.8

11. Post Hoc Outcome: Median Progression Free Survival
Description: as for outcome 2
Time Frame: From the start of treatment and every 2 cycles, where 1 cycle equals 28 days, during treatment. Median follow up at time of data was 33 months.
Population: Two patients were not evaluable
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
Number analyzed (Participants) | 46
months | 9.2 [6.4 to 11.3]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected over a 9 year period for the study. AEs were assessed and recorded at the beginning of each cycle (1 cycle =28 days) while on treatment and 30 days beyond the last treatment for a maximum of 69 cycles (the most number of cycles any patient was treated on study)
Arm/Group | Erlotinib and Bevacizumab Combination Treatment
All-Cause Mortality (participants affected / at risk) | 43/48
Serious Adverse Events (participants affected / at risk) | 15/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Bevacizumab Combination Treatment (N=48)
Hypertension (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Small bowel perforation (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Death (Injury, poisoning and procedural complications) | 1 (1)
International Normalized Ratio of Prothrombin time (INR) (Injury, poisoning and procedural complications) | 1 (1)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Potassium - serum low (Metabolism and nutrition disorders) | 1 (1)
General Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Facial droop (Nervous system disorders) | 1 (1)
Neuropathy - Motor (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound complication (non infectious) (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib and Bevacizumab Combination Treatment (N=48)
Allergic rhinitis (Immune system disorders) | 6
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 10
Leukocytes (total white blood cells) (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 25
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 10
Hypertension (Cardiac disorders) | 12
Sinus bradycardia (Cardiac disorders) | 3
Fatigue (General disorders) | 29
Fever (General disorders) | 3
Insomnia (General disorders) | 4
Rigors (General disorders) | 5
Weight loss (General disorders) | 11
Brusing (Skin and subcutaneous tissue disorders) | 5
Cheilitis (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 16
Nail changes (Skin and subcutaneous tissue disorders) | 7
Pruirtus/itching (Skin and subcutaneous tissue disorders) | 18
Rash acne (Skin and subcutaneous tissue disorders) | 13
Rash/desquamation (Skin and subcutaneous tissue disorders) | 36
Anorexia (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 11
Dehydration (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 39
Dry mouth (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 4
Heartburn (Gastrointestinal disorders) | 7
Hemorrhoids (Gastrointestinal disorders) | 10
Incontinence anal (Gastrointestinal disorders) | 3
Mucositis/stomatitis (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 24
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 9
Hemmorhage, GI rectum (Gastrointestinal disorders) | 5
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 11
Petechiae/purpura (Skin and subcutaneous tissue disorders) | 4
Sinus infection (Infections and infestations) | 4
Upper airway infection (Respiratory, thoracic and mediastinal disorders) | 3
Urinary tract infection (Infections and infestations) | 6
Skin rash (Infections and infestations) | 3
Edema in limbs (Blood and lymphatic system disorders) | 7
Albumin - serum low (Metabolism and nutrition disorders) | 19
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Serum glutamic pyruvic transaminase (ALT/SGPT) (Metabolism and nutrition disorders) | 7
serum glutamic oxaloacetic transaminase (AST/SGOT) (Metabolism and nutrition disorders) | 11
Bicarbonate - serum low (Metabolism and nutrition disorders) | 3
Bilirubin, serum high (Metabolism and nutrition disorders) | 22
Calcium, serum low (Metabolism and nutrition disorders) | 8
Creatinine, high (Metabolism and nutrition disorders) | 6
Glucose, serum high (Metabolism and nutrition disorders) | 19
Glucose, serum low (Metabolism and nutrition disorders) | 8
Lactic acid dehydrogenase (LDH) (Metabolism and nutrition disorders) | 5
Magnesium, serum low (Metabolism and nutrition disorders) | 15
Phosphate, serum high (Metabolism and nutrition disorders) | 3
Phosphate, serum low (Metabolism and nutrition disorders) | 4
Potassium, serum high (Metabolism and nutrition disorders) | 8
Potassium, serum low (Metabolism and nutrition disorders) | 11
Proteinuria (Metabolism and nutrition disorders) | 6
Sodium, serum high (Metabolism and nutrition disorders) | 7
Decreased Uric acid (Metabolism and nutrition disorders) | 3
Chloride, serum high (Metabolism and nutrition disorders) | 4
Carbon dioxide increased (Metabolism and nutrition disorders) | 6
Protein - decreased (Metabolism and nutrition disorders) | 4
Increased Blood Urea Nitrogen (BUN) (Metabolism and nutrition disorders) | 6
Extremity lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 9
Joint function (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness, generalized or specific area - lower extremity (Musculoskeletal and connective tissue disorders) | 6
Muscle weakness, generalized or specific area - whole body (Musculoskeletal and connective tissue disorders) | 7
Ataxia (incoordination) (Nervous system disorders) | 3
Cognitive disturbance (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Confusion (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 12
Memory impairment (Nervous system disorders) | 12
Mood alteration - Agitation (Psychiatric disorders) | 5
Mood alteration - Anxiety (Psychiatric disorders) | 5
Mood alteration - Depression (Psychiatric disorders) | 9
Sensory Neuropathy (Nervous system disorders) | 5
Pyramidal tract dysfunction (increased tone, hyperreflexia, positive Babinski, decreased fine motor) (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 7
Speech impairment (e.g. dysphasia/ aphasia) (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 5
Dry eye syndrome (Eye disorders) | 6
Vision impairment (hemianopsia/quadrantanopia) (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 6
Extremity- limb pain (Musculoskeletal and connective tissue disorders) | 8
Joint pain (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 23
Throat pain (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria ( hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 5
Urinary incontinence (Renal and urinary disorders) | 4
Thrombosis/embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No